CLINICAL TRIAL: NCT00928122
Title: Intrastromal Correction of Ametropia by a Femtosecond Laser
Acronym: ISCAF
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: 20/10 Perfect Vision (Industry)
Responsible Party: Priv.-Doz. Dr. med. Mike P. Holzer, Universitaets-Augenklinik Heidelberg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISCAF
Record Dates: First submitted 2009-06-03; First posted 2009-06-25 (Estimated); Last update posted 2010-02-09 (Estimated); Status verified 2010-02

CONDITIONS: Presbyopia; Myopia; Hyperopia; Astigmatism
MeSH Terms: conditions — Presbyopia; Myopia; Hyperopia; Astigmatism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 / Presbyopia (Experimental): Presbyopic patients, slightly hyperopes
  Interventions: Device: Intrastromal Correction of Presbyopia
- 2 / Myopia (Experimental): Myopic patients without Astigmatism
  Interventions: Device: Intrastromal correction of Myopia
- 3 / Hyperopia (Experimental): Hyperope patients without Astigmatism
  Interventions: Device: Intrastromal Correction of Hyperopia
- 4 / Myopia with Astigmatism (Experimental): Myopic patients incl. Astigmatism
  Interventions: Device: Intrastromal Correction of Myopia incl. Astigmatism
- 5 / Hyperopia with Astigmatism (Experimental): Hyperope patients incl. Astigmatism
  Interventions: Device: Intrastromal Correction of Hyperopia incl. Astigmatism

INTERVENTIONS:
Device: Intrastromal Correction of Presbyopia — Applying defined, pre-programmed patterns (e.g. rings and/or radial cuts)into the human eye cornea. It is a minimal-invasive procedure which changes the topography of the cornea and by that the refraction ability.
  Other Names: - FEMTEC Laser System; - Patient Interface
  Arms: 1 / Presbyopia
Device: Intrastromal correction of Myopia — Applying defined, pre-programmed patterns (e.g. rings and/or radial cuts)into the human eye cornea. It is a minimal-invasive procedure which changes the topography of the cornea and by that the refraction ability.
  Other Names: FEMTEC Laser System
  Arms: 2 / Myopia
Device: Intrastromal Correction of Hyperopia — Applying defined, pre-programmed patterns (e.g. rings and/or radial cuts)into the human eye cornea. It is a minimal-invasive procedure which changes the topography of the cornea and by that the refraction ability.
  Other Names: FEMTEC Laser System
  Arms: 3 / Hyperopia
Device: Intrastromal Correction of Myopia incl. Astigmatism — Applying defined, pre-programmed patterns (e.g. rings and/or radial cuts)into the human eye cornea. It is a minimal-invasive procedure which changes the topography of the cornea and by that the refraction ability.
  Other Names: FEMTEC Laser System
  Arms: 4 / Myopia with Astigmatism
Device: Intrastromal Correction of Hyperopia incl. Astigmatism — Applying defined, pre-programmed patterns (e.g. rings and/or radial cuts)into the human eye cornea. It is a minimal-invasive procedure which changes the topography of the cornea and by that the refraction ability.
  Other Names: FEMTEC Laser System
  Arms: 5 / Hyperopia with Astigmatism

SUMMARY:
This study evaluates the intrastromal correction of ametropia with a femtosecond laser made by 20/10 PERFECT VISION. This laser generates a beam of ultrashort, infrared pulses which enables very precise cuts in the cornea. By these cuts lamellae of the cornea are separated locally, and in the consequence the curvature of the cornea is changed, and the correction of the diagnosed ametropia can be achieved. On the contrary to cuts which are generated with a sharp knife, the cuts generated when using a laser can be generated just inside the cornea without opening the surface of the cornea. This means the procedure is minimal-invasive.

The study hypothesis is: Different types of ametropia can be corrected safely and on long-term by intrastromal cuts.

ELIGIBILITY:
Inclusion Criteria:

* age: > 18 years
* stable distance refraction for at least one year (i.e. a maximum change of 0.5 D)
* in the case of presbyopia: minimum near add +2D to + 4D
* in the case of myopia or hyperopia (without astigmatism): minimal 1D and maximum 3D
* in the case of myopia or hyperopia (with astigmatism): spherical equivalent of minimal 1D and maximum 3D
* BSCVA of the eye to be treated >= 0.63
* patients are willing and in such conditions to come to the follow-up exams
* no further ocular pathologies

Exclusion Criteria:

* age: < 18 years
* refraction less than +/- 1 D or higher than +/- 3 D (not valid for presbyopia patients)
* minimal pachymetry of < 500µm
* K-mean < 37 D or > 60 D
* Difference (K-max minus K-min) > 5D
* Difference cycloplegic refraction to subjective refraction more than 1 D (valid only for hyperopia correction)
* patients with previous intraocular or corneal surgeries (e.g. post-LASIK or PRK patients). Exemption: standard cataract surgery.
* patients with one or more of the following ocular pathologies:

  * keratokonus
  * corneal scars
  * transplanted cornea
  * disorders of wound healing
  * trauma
  * glaucoma
  * epilepsia
  * nystagmus
  * lack of concentration
  * other complicated illnesses
  * diabetes mellitus
  * instable K-readings as a sign of instable cornea
  * weakness of connective tissue
  * sensitivity against the drugs used in the study
  * continuous wearing of contact lenses before the pre-exam, and before the surgery. At least 14 days before these dates patients must abstain from wearing CL.
  * patients in pregnancy or during lactation
  * patients who take part in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2008-07; Primary Completion 2009-01 (Actual); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Prove safety and effectiveness as well as improvement in near visual acuity performance and increase in near visual acuity. | 3 months

SECONDARY OUTCOMES:
Validate the 3 months results | 6 months
Prove stability of distance visual acuity and safety of the procedure regarding infections and inflammatory response as well as corneal endothelial cell counts. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Gerd U. Auffarth, Prof. Dr., Principal Investigator — Universitäts-Augenklinik Heidelberg
Locations (3):
- Germany (3):
  - Klinik für Refraktive und Ophthalmo-Chirurgie des EJK Niederrhein, Duisburg
  - FreeVis LASIK Zentrum Mannheim GmbH, Mannheim
  - Augenklinik am Marienplatz AG & Co. KG, München

REFERENCES:
- [Derived] Khoramnia R, Fitting A, Rabsilber TM, Thomas BC, Auffarth GU, Holzer MP. Intrastromal femtosecond laser surgical compensation of presbyopia with six intrastromal ring cuts: 3-year results. Br J Ophthalmol. 2015 Feb;99(2):170-6. doi: 10.1136/bjophthalmol-2014-305642. Epub 2014 Sep 2. PMID 25185255